CLINICAL TRIAL: NCT01288157
Title: A Randomized, Open-label Study to Evaluate the Pharmacokinetics of a Single Subcutaneous Administration of 50 mg or 100 mg Golimumab in a Pre-filled Syringe Formulation to Healthy Male Chinese Subjects
Brief Title: A Study of the Pharmacokinetics of Golimumab in Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016273; C0524T30
Record Dates: First submitted 2010-11-22; First posted 2011-02-02 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Healthy Adult Chinese Males
Keywords: healthy; adult; Chinese; male; Simponi; CNTO 148
MeSH Terms: interventions — golimumab

ARMS (2):
- 001 (Experimental): Golimumab Single dose of 50 mg subcutaneously
  Interventions: Drug: Golimumab
- 002 (Experimental): Golimumab Single dose of 100 mg subcutaneously
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Golimumab — Single dose of 100 mg subcutaneously
  Arms: 002
Drug: Golimumab — Single dose of 50 mg subcutaneously
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of golimumab in Chinese male participants.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned by chance), open-label (both the physician and subject know the assigned study medication) study to assess the safety, tolerability, immune response, pharmacokinetics (what the body does to the drug), of golimumab (Simponi). The study population will consist of 24 healthy male participants in China. Subjects will receive a single dose of either 50 mg or 100 mg golimumab. Subjects will be in the study for up to 14 weeks. Safety assessments will be performed throughout the study and include obtaining and evaluating laboratory tests, vital signs (eg, blood pressure), and the occurrence and severity of adverse events. A single dose of 50 mg or 100 mg golimumab as a subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

* Have no clinically relevant abnormalities
* non-smoker or agree to smoke no more than 10 cigarettes or 2 cigars per day throughout the study.

Exclusion Criteria:

* Have or had a history of clinically significant, severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease
* Have any underlying physical or psychological medical condition
* Be unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access to veins.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (area under the plasma concentration versus time curve [AUC] and Peak Plasma Concentration [Cmax]) of golimumab in Chinese male subjects | Day 71 (Week 11)

SECONDARY OUTCOMES:
Number of participants with adverse events | Day 71
Immunogenicity of golimumab, as measured by antibodies to golimumab | Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (1):
- Beijing, China